CLINICAL TRIAL: NCT00589511
Title: Nucleus Freedom Cochlear Implant System Pediatric Post-approval Study
Status: Completed | Type: Observational
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Other Study IDs: CORP5183
Record Dates: First submitted 2007-12-23; First posted 2008-01-09 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Sensorineural Hearing Loss
Keywords: Bilateral severe to profound sensorineural hearing loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Case-Only

SUMMARY:
The objective of this multisite study is to evaluate the performance of the Nucleus Freedom cochlear implant system in a large population of sequentially implanted pediatric subjects.

DETAILED DESCRIPTION:
The proposed study will include 50 pediatric subjects ages 1 year to 17 years, 11 months of age, implanted at up to 5 sites in the United States and Canada. The estimated duration of this multisite study is 18 to 24 months. The duration of individual subject participation is not to exceed 12 months.

The study will be conducted as a within-subject repeated measures experiment (in which each subject serves as his or her own control) in order to accommodate the heterogeneity that is well known to characterize hearing-impaired populations

ELIGIBILITY:
Inclusion Criteria:

* 1 year to 17 years, 11 months of age.
* Bilateral severe to profound sensorineural hearing loss for those 1 to 2 years of age. Severe hearing loss for those 2 years of age and older.
* Limited benefit from bilateral hearing aids. Limited benefit is defined as a lack of progress in the development of simple auditory skills in conjunction with appropriate amplification and intensive aural rehabilitation over a 3 to 6 month period.

  * For younger children, unable to take speech perception tests due to age-related cognitive and linguistic limitations, limited benefit will be quantified using the Infant Toddler Meaningful Auditory Integration Scale (IT-MAIS)1 or Meaningful Auditory Integration Scale (MAIS)1.
  * For older children, capable of speech perception tasks, limited benefit is defined as £ 30% on the recorded open-set Multisyllabic Lexical Neighborhood Test (MLNT)2 or Lexical Neighborhood Test (LNT) 2, depending on the child's cognitive and linguistic skills.
* English spoken as a primary language.
* Willingness to participate in and to comply with all requirements of the protocol.

Exclusion Criteria:

* Ossification or any other cochlear anomaly that might prevent complete insertion of the electrode array, as confirmed by medical examination and tests including MRI.
* Signs of retrocochlear or central origin to hearing impairment as confirmed by medical examination and tests including MRI.
* Medical or psychological conditions that would contraindicate undergoing surgery (e.g., active middle ear infections, tympanic membrane perforation).
* Additional handicaps that would prevent or restrict participation in the evaluations.
* Unrealistic expectations on the part of the subject or subject's parents/guardians, regarding the possible benefits, risks and limitations that are inherent to the surgical procedure and prosthetic device.
* Unwillingness or inability of the candidate or candidate's parents/guardians to comply with all study requirements.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with bilateral severe to profound sensorineural hearing loss who undergo implantation with the Nucleus Freedom Cochlear Implant System
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2006-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
IT-MAIS | 12 Months
MAIS | 12 Months
MLNT | 12 Months
LNT | 12 Months